CLINICAL TRIAL: NCT06489535
Title: Retention and Re-Engagement in Treatment for Addiction Following Serious Injection Related Infections (RETAIN): A Pilot Randomized Controlled Study
Brief Title: Retention and Re-Engagement in Treatment for Addiction Following Serious Injection Related Infections (RETAIN)
Acronym: RETAIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-44905; K23DA054363 (NIH)
Record Dates: First submitted 2024-06-28; First posted 2024-07-08 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Opioid Use Disorder; Bloodstream Infection; Osteomyelitis; Endocarditis; Septic Arthritis; Epidural Abscess
Keywords: Recovery Management Checkups (RMC); Serious injection related infections (SIRI); Medications for OUD (MOUD); Re-hospitalizations
MeSH Terms: conditions — Opioid-Related Disorders; Sepsis; Osteomyelitis; Endocarditis; Arthritis, Infectious; Epidural Abscess

STUDY DESIGN:
Intervention Model Description: The randomization process will involve assigning participants to either the intervention or control group The Randomization ratio will be 2:1 to intervention and will be done after enrollment by a research assistant through an automated Redcap feature.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RETAIN intervention (Experimental): Participants randomized to the RETAIN intervention will receive Motivational Interviewing targeted to their clinical concerns and personalized support tailored to each participants' specific needs determined by their answers to intake questions.
  Interventions: Other: RETAIN
- Control (Active Comparator): Control arm participants will be offered different videos or podcast episodes that are unrelated to the study topics of infections, substance use, overdose, and medication management.
  Interventions: Other: Unrelated videos

INTERVENTIONS:
Other: RETAIN — There are 6 different modules that a participant in the RETAIN intervention group can be placed in: "Reinforce Antibiotic Completion", "Linkage to Antibiotic Treatment/Alternate Plan", "Reinforce Recovery", "Linkage to MOUD/Alternate Plan", "Reinforce Treatment Attendance", and "Harm Reduction Support". Participants may be assigned to no more than three modules at a time until they finish their antibiotics. After the completion of antibiotics, participants may only be in two modules. Participants' intervention can range from 15 minutes- 60 minutes depending on what modules they are placed in and how much support they feel they need. Interventions will begin at the two-week follow up after a participant has been discharged from Boston Medical Center (BMC).
  Arms: RETAIN intervention
Other: Unrelated videos — These videos unrelated to the study topics will last approximately 30-45 minutes. Depending on the method of communication, participants will watch a video (in person) or listen to a podcast (remote)
  Arms: Control

SUMMARY:
This project is a pilot study of an adapted intervention of an existing Opioid Use Disorder (OUD) treatment retention intervention called Recovery Management Checkups (RMC). This intervention has been adapted to better fit the experiences and unique issues of those that have been hospitalized with serious injection related infections (SIRI) based on the findings from a prior qualitative study from the principal investigator. This project plans to test the adapted intervention within a smaller group of participants to assess feasibility, acceptability, and calculate early findings of intervention efficacy.

Hospitalizations for SIRIs are a unique entry point for patients to start their recovery journey with medications for OUD (MOUD), but many people do not remain on long-term treatment, despite evidence that indicates MOUDs reduce death and re-hospitalization after SIRIs.

The study objectives are to:

* Assess the implementation feasibility of the adapted RMC model for patients with SIRI and OUD.
* Establish preliminary estimates of intervention efficacy.
* Make further adaptions to the intervention that will reduce both known and unknown barriers to care and increase effectiveness in future larger scale trials.

Findings from this pilot study will result in further intervention refinement to better fit the target population, and serve as the basis for a larger randomized control trial that will have aims focused on more in-depth analysis of the efficacy of this program

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 65 years of age
* Able to provide Informed Consent
* Admitted to Boston Medical Center on any inpatient unit for an active serious injection related infection (SIRI) such as endocarditis, osteomyelitis, bacteremia, septic arthritis, epidural abscess or other serious infection in which two weeks or more of antibiotics are recommended

Exclusion Criteria:

* Not able to give informed consent
* Cognitive ability (defined through Research Assistant (RA) determination)
* Inability to complete assessments in English or Spanish (defined through RA determination).
* Exclusion for any reason under PI discretion
* Unable to provide names and contact information for at least two verifiable locator persons who will know where to find them in the future.
* In police custody or expecting incarceration

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of days on medications for opioid disorder (MOUD) | Baseline while hospitalized, then 2 weeks, 6 weeks, 3 months, and 6 months after discharge
  The timeline follow back (TLFB) method will be used to assess this outcome based on self-report.
Participant recruitment rates | Baseline while hospitalized, then 2 weeks, 6 weeks, 3 months, and 6 months after discharge
  Participant recruitment rates will be calculated by dividing the number of participants enrolled by the number of eligible patients identified.
Feasibility of the RETAIN Intervention based on completion of study visits | Baseline while hospitalized, then 2 weeks, 6 weeks, 3 months, and 6 months after discharge
  The rates of completion of study visits will be calculated by dividing the number of completed study visits by the total number of study visits.
Acceptability of the RETAIN Intervention | Baseline while hospitalized, then 2 weeks, 6 weeks, 3 months, and 6 months after discharge
  Acceptability will be assessed using the Acceptability of Intervention Measure (AIM) which is a 4-item measure of perceived intervention acceptability. Items are measured on a 5-point Likert scale (Completely Disagree-Completely Agree). Score is calculated mean and higher scores are associated with better acceptability.

SECONDARY OUTCOMES:
Number of days of antibiotic completion | Baseline while hospitalized, then 2 weeks, 6 weeks, 3 months, and 6 months after discharge
  Self-report yes or no.
Number of days of Opioid use | Baseline while hospitalized, then 2 weeks, 6 weeks, 3 months, and 6 months after discharge
  The TLFB method will be used to assess this outcome based on self-report.
Number of Hospitalizations | Baseline while hospitalized, then 2 weeks, 6 weeks, 3 months, and 6 months after discharge
  The TLFB method will be used to assess this outcome based on self-report.
Number of uncleaned injections | Baseline while hospitalized, then 2 weeks, 6 weeks, 3 months, and 6 months after discharge
  Self Report based on the The Bacterial Skin Index Risk Score (BIRSI) score, which includes questions about alcohol pad and sterile water use, handwashing, rotating injection sites, injecting subcutaneously or in the muscle ("skin/muscle popping"), and clean needle use, was used as a continuous score to measure risk of skin and soft tissue infections.
Number of unmonitored opioid use | Baseline while hospitalized, then 2 weeks, 6 weeks, 3 months, and 6 months after discharge
  Self Report based on Opioid use
MOUD stigma | Baseline while hospitalized, and 6 month after discharge
  Partial adaptation of MMT-SMS stigma scale will be used to assess this outcome based on self-report

CONTACTS AND LOCATIONS:
Overall Officials: Simeon Kimmel, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No